CLINICAL TRIAL: NCT01140763
Title: Tissue Sampling Bias in Histologic Evaluation of Sentinel Lymph Nodes in Breast Cancer
Brief Title: Clinical Evaluation of Tissue Sampling Bias in Histologic Evaluation of Sentinel Lymph Nodes in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sysmex America, Inc. (Industry)
Responsible Party: Carrie Pineda, Sysmex America, Inc
Other Study IDs: Histo-BC-001
Record Dates: First submitted 2010-06-03; First posted 2010-06-09 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Breast Neoplasms; Breast Diseases
Keywords: metastasis
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sysmex's 5-blade cutter.
  Interventions: Device: Sysmex's 5-blade lymph node cutter

INTERVENTIONS:
Device: Sysmex's 5-blade lymph node cutter — A maximum of 3 dissected sentinel lymph nodes (SLN) per subject will be included in this study. Lymph nodes will be sliced at 1 mm intervals with Sysmex's 5-blade lymph node cutter. Alternate slices will be allocated to either "reference" histopathology or "test" histopathology. Three serial sections will be cut every 200 µm (level): the 1st section per level for hematoxylin & eosin (H&E), the middle section of the 3rd level for Immunohistochemistry (IHC)(pan- cytokeratin antibody clone AE1/AE3). All other sections will be blanks in case further analysis is needed.

SUMMARY:
This is a study to evaluate the incidence of sampling bias during pathologic assessment of sentinel lymph nodes (SLN) when they are cut at a certain thickness (1 mm) and the tissue slices are completely analyzed by histopathology (at 200 µm sections). The sponsor and investigators would like to determine how often small cancer deposits are present in one slice but not the other. The data will provide an empirical estimate of the incidence of tissue sampling bias inherent in using different tissue sections for analysis. The data will also show how varying degrees of detail in evaluating the sentinel lymph nodes (SLN) with histopathology methods will impact the degree of agreement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Diagnosed pre-surgically with T1 or T2 breast cancer and scheduled for surgery including sentinel lymph node dissection
* Subjects (or the subject's legal representative) who have read, understood (to the best of their ability) and signed the informed consent form.

Exclusion Criteria:

* Subjects diagnosed pre-surgically with large or locally advanced (T3 & T4) breast cancer
* Pregnant subjects, confirmed by interview with either subject or treating physician
* Subjects diagnosed with inflammatory breast cancer
* Subjects diagnosed with ductal carcinoma in situ (DCIS) when breast conservation is to be done
* Subjects with clinically suspicious, palpable axillary lymph nodes
* Subjects previously treated for or previously diagnosed with another type of invasive cancer. Subjects with skin cancer (basal cell and squamous cell carcinoma) may be included, except for subjects diagnosed with melanoma
* Subjects who have received pre-operative systemic therapy
* Subjects who are incapable of providing written informed consent
* Subjects who have been judged to be an inappropriate candidate by any medical care provider (e.g., surgeon, oncologist or pathologist).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a previous diagnosis of breast cancer scheduled for sentinel lymph node dissection.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Prospectively assess the agreement of histopathology results on tissue sections taken from different slices of SLNs removed using standard SLN biopsy procedures. | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Care Specialist, PC, Allentown, Pennsylvania, United States